CLINICAL TRIAL: NCT04200131
Title: Histological Diagnostic Value of the Moray Micro Forceps in the Management of Pancreatic Cysts.
Brief Title: Moray Micro Forceps and Pancreatic Cyst
Acronym: MOBIDYC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VANBIERVLIET (Other)
Responsible Party: Sponsor-Investigator, VANBIERVLIET, Director, Head of Endocopy, Principal Investigator, Medical doctor, Société Française d'Endoscopie Digestive
Organization: Société Française d'Endoscopie Digestive (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SFED N 133
Record Dates: First submitted 2019-12-03; First posted 2019-12-16 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pancreas Cyst
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moray micro-forceps (Experimental)
  Interventions: Diagnostic Test: Biopsy of the cyst wall with the Moray™ forceps.

INTERVENTIONS:
Diagnostic Test: Biopsy of the cyst wall with the Moray™ forceps. — Tissue sample of the wall of the pancreatic cyst with micro Moray™ forceps during an ultrasound-guided puncture of a pancreatic cyst with a 19G needle.

SUMMARY:
The prevalence of pancreatic cysts in the general population is high close to 1%. The diagnosis is most of the time fortuitous thanks to the improvement of the imaging resources available. These lesions include a large number of entities, some of with malignant potential. Mucinous lesions present a high risk of tumor transformation, justifying surgery, which is sometimes heavy. It appears essential to select the best patients to benefit from this type of treatment. For this purpose, the accuracy of the diagnostic means must be optimal. The Fine Needle Aspiration under Endoscopic ultrasound, validated in this context, have a low complication rate. It allows a cytological evaluation and analysis of tumor markers measurements in cystic fluid. However, cytopathological evaluation is only contributing in 1/3 to half of cases. The assays of markers (including the main one ACE) have high specificities but high insufficient sensitivities (less than 50%). Molecular techniques (K-RAS mutation in particular), of variable availability, allow to increase the sensitivity in association with the other diagnostic parameters. But the rate of false negatives remains above 20% to date. A diagnostic means to obtain a histology of the cyst wall would reduce considerably the risk of error.

The Moray™ micro forceps is forceps that aims to provide a tissue sample of the wall of the pancreatic cyst. It is inserted into a commonly used 19 Gauge needle during the puncture of the cyst under endoscopic ultrasound. It could increase the accuracy diagnosis of the procedure. These forceps has recently become available to the practitioner and has obtained the CE marking.

To date, no quality multi-center prospective evaluation has determined the capacity of to obtain a histology of the pancreatic cystic walls by this technique. Its safety must be also be accurately assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* FNA of the cystic fluid indicated during an endoscopic ultrasound examination
* Abdominal CT and pancreatic MRI less than 3 months old, available
* Pancreatic cyst unilocular or with a macrolocule in case of multilocular cyst, of size ≥ to 20 mm of major axis with a clean wall.

Exclusion Criteria:

* Contraindication to performing an upper endoscopic ultrasound
* Patient with known chronic calcifying pancreatitis, or suspected on the iconography available during the screening visit
* Patient taking an antiplatelet, or anticoagulant therapy including anti-vitamin K, direct oral anticoagulant, or heparin.
* Hemorrhagic disease, hemostasis and coagulation disorder (TP < 60%, TCA > 40 sec. and platelets < 60000/mm3), malignant hematopathy, chronic cirrhotic liver disease with Child Pugh B or C, acute or severe chronic renal failure (creatinine clearance < to 30 ml/min)
* Mental disability of the subject making participation in the trial impossible
* Patient not affiliated to a social security system
* Inability to understand or sign informed consent
* Serious adverse events
* Early termination of participation, withdrawal of voluntary informed consent of the patient
* Violation of protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Obtaining histological diagnosis by using "The Moray" micro forceps. | Day 10
  Obtaining enough tissue material by using "The Moray" micro forceps allowing paraffin embedding, histological analysis and diagnosis according to the opinion of the pathologist. The ability of the micro-forceps to obtain a positive sample will be determined histologically. The proportion % of the positive samples (diagnosis from the pathologist) will correspond to the number of patients whose histological diagnosis is obtained according to the pathologist (tissue with presence of a chorion / extracellular matrix) divided by the total number of patients enrolled in this trial.

SECONDARY OUTCOMES:
The diagnostic accuracy of the technique (The Moray" micro forceps) | 6 months
  The diagnostic accuracy of the technique will be determinate by comparison between the results obtained after using the Moray micro forceps and diagnosis retained after surgery. If the surgery is not performed, the diagnostic accuracy will be determined by 3 independent experts by using the morphological results of the different iconographies, cytology, intracystic fluid dosages
Emergent Adverse Events of the technique (the Moray micro-forceps) | Day 0 and after 1 month
  The emergent adverse events will be assessed (Moray micro forceps) by compilation of all adverse events occurring immediately or at 30 days post-procedure (hemorrhages, possible episodes of acute pancreatitis or infection) according to degree of the severity: slight, moderate, severity, and fatal( cotton's criterions).The proportion of patients presenting at least one morbid event during the biopsy and after post-procedure (immediately) will be calculated and compared by using Prescott test. In the same way, the delayed morbidity of the procedure as a whole will be described by the proportion of patients who had a morbid event delayed between the end of the procedure and Day 30.
Technical success of the Moray micro-forceps | Day 0
  Assessed by the proportion of patients whose procedure allow obtained a biopsy in absence of a technical incident: passage of the micro-forceps through the 19G needle, its opening, the acquisition of tissue material, and its removal from the needle at the end of the procedure.
Satisfaction of the technique (Moray micro-forceps) on the management of pancreatic cyst | 6 months
  Estimated by the proportion of patients for which the decision by the monitoring experts was different after obtaining the result of the samples by the Moray micro-forceps compared to a usual support based on the techniques available today.
Quality of the sample | Day 10
  Determined by the proportion of samples with a histological analyzable surface by the pathologist.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Archet II, Nice, France